CLINICAL TRIAL: NCT06942728
Title: Personalized Medicine in the Elderly With Vision Impairment and Mild Cognitive Impairment: Effects of Sensorineural Telerahabilitation
Brief Title: Personalized Medicine in the Elderly With Vision Impairment and Mild Cognitive Impairment
Acronym: Eye-MCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5032
Record Dates: First submitted 2025-03-24; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sperimental (Experimental): All patients will undergo:
  * Standardized battery of tests for the diagnosis of cognitive decline corresponding to the BDM (Battery for Mental Deterioration
  * Global assessment measure of cognitive status (Minimal Mental State Examination - MMSE)
  * Complete eye examination
  * Tonometry
  * Visual acuity for distance (ETDRS) and near (MNRead)
  * Reading speed (IrestTEST)
  * Microperimetry
  * Psychological evaluation
  * Patients with visual impairment randomized to receive neurovisual rehabilitation treatment will carry out neurosensory rehabilitation remotely.
  Interventions: Device: nLIFE EyeFitness
- Control (No Intervention): All patients will undergo:
  * Standardized battery of tests for the diagnosis of cognitive decline corresponding to the BDM (Battery for Mental Deterioration
  * Global assessment measure of cognitive status (Minimal Mental State Examination - MMSE)
  * Complete eye examination
  * Tonometry
  * Visual acuity for distance (ETDRS) and near (MNRead)
  * Reading speed (IrestTEST)
  * Microperimetry
  * Psychological evaluation

INTERVENTIONS:
Device: nLIFE EyeFitness — A software called nLIFE EyeFitness, certified as a Class I Medical device, allows to carry out individualized rehabilitation exercises at home, using own PC or tablet, with monitoring by the Center's operators.
  Arms: Sperimental

SUMMARY:
Globally, approximately 55 million people suffer from dementia, and 60-70% of cases are due to Alzheimer's disease (AD). Increasing scientific evidence highlights that the pathological changes underlying AD and other forms of dementia begin long before the onset of symptoms. Mild cognitive impairment (MCI) is a clinical condition that in people over 65 shows a prevalence ranging from 3% to 22%. The characteristics of MCI are the presence of a subjective memory disorder and a reduced ability to learn new information with normal general cognitive functioning, normal ability to perform daily activities and the absence of other conditions, such as depression, that could justify the memory disorder. Currently, the diagnosis of MCI is based exclusively on clinical evaluation, including neuropsychological tests.

Currently, there are no therapies available to prevent and/or treat dementia and the options for intervention are represented by treatments such as physical exercise and cognitive treatment. These practices refer to the concept of cognitive reserve. Computerized cognitive training (CCT) is characterized by being a personalized intervention, allows multi-domain training and increases the cognitive processes of patients with MCI. The National Low Vision Center has been using a software called nLIFE EyeFitness for several years, certified as a Class I Medical device. It allows you to carry out individualized rehabilitation exercises at home, using your own PC or tablet, with monitoring by the Center's operators. The exercises currently present stimulate attention, short-term visual memory, reaction time, executive function, working memory and, therefore, also appear suitable for stimulating subjects with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 60 years with a diagnosis of aMCI
* Signing of informed consent

Exclusion Criteria:

* Age <60 years
* History of dementia
* Diabetes mellitus
* Uncontrolled hypertension
* Diagnosis of major depression
* Glaucoma
* Age-related macular degeneration
* Media opacity and vitreoretinal pathologies that may preclude a correct evaluation
* • Failure to obtain informed consent

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The effects of neurosensory telerehabilitation in elderly subjects with MCI | 8 months
  Evaluate the effects of neurosensory telerehabilitation in terms of reduction of cognitive deterioration by evaluating the scores of neuropsychological questionnaires in use in clinical practice after using the remote neurovisual rehabilitation platform in use at the Polo Nazionale di Ipovisione

SECONDARY OUTCOMES:
Evaluation the effects of neurosensory telerehabilitation on visual tests score | 8 months
  Evaluate the effects of neurosensory telerehabilitation, in terms of variation in visual test scores, in elderly subjects affected by visual impairment and MCI using the remote neurovisual rehabilitation platform in use at the Polo Nazionale di Ipovisione.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Turco, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Polo Nazionale Ipovisione, Rome, Lazio, Italy